CLINICAL TRIAL: NCT03142997
Title: Effect of Spontaneous Ventilation Versus Controlled Ventilation on Lung Atelectasis Assessed by Lung Ultrasound in Children.
Brief Title: Spontaneous Ventilation Versus Controlled Ventilation on Lung Atelectasis in Children.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Lotfy, Principle investigator, Lecturer of anesthesia and intensive care, Cairo University
Other Study IDs: N-24-2017
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Lung Collapse
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group S: anesthetized children on spontaneous ventilation.
  Interventions: Diagnostic Test: Lung ultrasound
- group C: anesthetized children on controlled ventilation.
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — we will perform lung ultrasound for both groups to calculate lung score.

SUMMARY:
This is an observational study to compare the effect of spontaneous ventilation versus controlled ventilation on lung atelectasis using lung score measured by lung ultrasound. the study will be conducted in children hospital of Cairo University Hospitals and study population will be : children aged from one to eight years of age. primary outcome will be the lung score measured by lung ultrasound.

DETAILED DESCRIPTION:
Randomization will be done by computer generated numbers and concealed by serially numbered,opague and sealed envelopes. The details of the series will be unknown to the investigators and the group assignment will be kept in asset of sealed envelopes each bearing only the case number on the outside. Prior to surgery the appropriate numbered envelopes will be opened by the nurse, the card inside will determine the patient group. All children will be premedicated with oral midazolam 0.5mg/kg half hour before procedure and atropine at a dose of 0.01-0.02 mg/kg (IM). Continuous electrocardiogram (ECG), pulse oximetry, non-invasive arterial blood pressure, and temperature monitoring will be applied and all patients will be induced with inhalational anesthetic using Sevoflurane+ oxygen (O2) with mac 6%. After deepening of the anesthesia, intravenous (I.V.) line will be inserted and fentanyl 1μg/kg. Patient will be divided into two groups; group S (spontaneous) will be intubated and maintained spontaneously with Ayres T piece circuit on isoflurane + oxygen with mac 2% and with fresh gas flow 2 times minute ventilation of patient to avoid co2 rebreathing . Group C (controlled) will receive muscle given in the form of atracurium 0.5mg/kg and patients will be intubated by appropriate size of endotracheal tube. Patients in controlled group will be ventilated at 6 ml/ kg tidal volume, Inspiratory to expiratory (I: E) ratio 1:2, Fio2 1 and PEEP 5 cmH2o.

10 minutes after induction lung ultrasound will be done to assess lung score and arterial blood gases will be withdrawn. At the end of surgery lung ultrasound (LUS) will be done again and another blood gases will be taken.

LUS will be performed with the portable echograph MicroMax (SonoSite, M-turbo) using a linear probe of 3 to 6 MHz. Each hemithorax will be divided into six sections using three longitudinal lines (parasternal, anterior, and posterior axillary) and two axial lines, one above the diaphragm and another one 1 cm above the nipples.

As LUS provides regional information, we will repeat the following examination sequence in each hemithorax and in all patients: (1) anterior, (2) lateral, and (3) posterior regions starting from the diaphragm (caudal lung) and moving toward the apex (cranial lung). Each hemithorax will be assessed using the two-dimensional classical view placing the probe parallel to the ribs .The LUS of a normal lung shows a lung sliding (caused by the respiratory movement of the visceral pleura relative to the fixed parietal pleura) and A lines (repetitive horizontal reverberation artifacts generated by air within the lungs separated by regular intervals, the distances of which being equal that between the skin and the pleural line).

The lung ultrasound (LUS) assessment will be segmented in anterior , lateral (L) and posterior (P) regions in both lungs. The dotted black axial line separated the lungs in superior and inferior portions. Ovals depicted where the probe is placed in the classical LUS approach: mid-clavicular, lateral and posterior axillary lines.

Anesthesia-induced atelectasis would be associated with the following LUS signs:

* Localized iso- or hypoechoic areas as compared with the highly reflective or anechoic normally aerated lung tissue.21-25 This consolidation or tissue-like pattern is caused by a loss of lung aeration. It commonly arises from the pleural line and thus can be described as Juxtapleural consolidations of various sizes.
* Static air bronchograms are observed as bright echogenic branching structures within these lung consolidations.
* The juxtapleural consolidations commonly erases the typical normal A lines and a few focal B lines (vertical, laser-like lines that erase normal A lines) can be observed below them.
* The lack of local respiratory movement or lung sliding and the presence of the pulse sign (a small motion within the lungs caused by the transmission of heart beats through the atelectatic area) are sometimes observed in large atelectatic areas.

Patients' demographic data will be collected; age, gender, weight, height, type of surgery and duration of surgery.

Lung ultrasound examinations will be performed at different time-points 10 minutes after induction of general anesthesia and before extubation to detect lung atelectasis. Arterial blood samples will be collected simultaneously to measure Pao2.

Atelectasis will be assessed by ultrasound using lung aeration score applied for each region. Lung score is four points (0 = normal lung, 1 = moderate aeration loss, 2 = severe aeration loss, 3 = complete aeration loss and consolidation) so, applying score for 12 regions bilateral will result in maximum score 36 and lowest score 0.

Assessment of postoperative pulmonary complications like; postoperative lung collapse, postoperative pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II
* Children undergoing minor surgeries in supine position.

Exclusion Criteria:

* Parents' refusal.
* Patients with congenital heart disease.
* Patients with chronic pulmonary disease ( asthma, bronchiectasis, emphysematous disease, etc.,)
* Patients with respiratory tract infection.
* Patients with chest wall deformities.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children undergoing anesthesia for non-major surgical procedures in Cairo Univesity children hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

PRIMARY OUTCOMES:
Arterial oxygen tension (Pao2) | 10 minutes following induction of general anesthesia

SECONDARY OUTCOMES:
The lung aeration score | 10 minutes following induction of general anesthesia
  lung ultrasound will be per formed on 6 areas on each hemi-thorax and the total score will be calculated (from 0-3 on each area, so the total will be 36 maximum).
Correlation between lung score and Pao2. | 10 minutes following induction of general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Children Hospital "Aborreesh", Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No